CLINICAL TRIAL: NCT05247099
Title: Constructing Children's Eye Data Sharing Platform in Multiple Centers and Multiple Disciplines
Brief Title: Pediatric Eye Care Investigated Team
Acronym: PECT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: Affiliated Foshan Maternity & Child Healthcare Hospital, Southern Medical University ( Foshan Maternity & Child Healthcare Hospital) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021KYPJ185
Record Dates: First submitted 2022-01-06; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-01

CONDITIONS: Eye Diseases; Ocular Surface Disease; Systemic Disease; Children
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with systemic diseases: Systemic diseases such as Nephritic syndrome, and other systemic diseases that can affect the eyes.
- healthy children: The exclusion criteria for the subjects were eye diseases or other systemic diseases that can affect the quality or volume of tears or the secretion of tears. These included
  1. eyelid diseases: eyelid entropion, eyelid ectropion, ptosis, and palpebral dyskinesia;
  2. conjunctival diseases: pterygium and conjunctivitis;
  3. history of ocular surface chemical injury;
  4. history of eye surgery within 6 months or history of retinal laser photocoagulation;
  5. systemic diseases: Sjogren syndrome, Parkinson's disease, rheumatoid arthritis, Grave's disease, systemic lupus erythematosus, and others.

SUMMARY:
Use cohort research to analyze and compare eyes of healthy children and children with systemic diseases. Understand and analyze the incidence, characteristics and influencing factors of children's ocular surface diseases. Establish a multi-center children's eye data sharing platform to provide basic data support for the diagnosis and treatment of children's ocular surface diseases.

DETAILED DESCRIPTION:
Use cohort research to analyze and compare eyes of healthy children and children with systemic diseases. Understand and analyze the incidence, characteristics and influencing factors of children's ocular surface diseases. Establish a multi-center children's eye data sharing platform to provide basic data support for the diagnosis and treatment of children's ocular surface diseases.

All participants will be recruited from Zhongshan Ophthalmic Center, Sun Yat-sen University and Affiliated Foshan Maternity & Child Healthcare Hospital, Southern Medical University. Only children with written informed consent from their parents can participate in this study.

Participants will be excluded for (1) age>18; (2) previous use of orthokeratology lenses or low-concentration atropine; (3) allergy to compound tropicamide eye drop; (4) any history of ocular surgery.

All participants will undergo optometry and biometric measurements by a trained team. The axial length (AL), central corneal thickness (CCT), anterior corneal radii of curvature, anterior chamber depth (ACD), lens thickness (LT), the curvature power of the central flat meridian (K1) and the central steep meridian (K2), the ocular surface and fundus will be measured. All measurements will be taken in room light condition (1000 lux).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age≤18
* 2. Cooperate with eye examination
* 3. Sign informed consent

Exclusion Criteria:

* 1. Cannot cooperate with eye examination
* 2. The researcher believes that the patient is not suitable to participate in the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Choose suitable patients from the ophthalmology hospital outpatient clinic or the ophthalmology and pediatric outpatient clinics of the Maternal and Child Health Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
change of the non-invasive tear break-up time | baseline, 24th months
  change of the non-invasive tear break-up time in seconds
change of the lipid layer of tear film | baseline, 24th months
  change of the lipid layer of tear film in nanometers

SECONDARY OUTCOMES:
vision | baseline, 6th months, 12th months, 18th months, 24th months
  spherical equivalent in diopters
intraocular pressure | baseline, 6th months, 12th months, 18th months, 24th months
  the intraocular pressure in mm Hg
Eye axis length | baseline, 6th months, 12th months, 18th months, 24th months
  Eye axis length in millimeters
Anterior chamber depth | baseline, 6th months, 12th months, 18th months, 24th months
  Anterior chamber depth in millimeters
central corneal thickness | baseline, 6th months, 12th months, 18th months, 24th months
  central corneal thickness in millimeters
Lens thickness | baseline, 6th months, 12th months, 18th months, 24th months
  Anterior chamber depth in millimeters
Retina thickness | baseline, 6th months, 12th months, 18th months, 24th months
  retina thickness in millimeters
choroid thickness | baseline, 6th months, 12th months, 18th months, 24th months
  choroid thickness in millimeters
Corneal curvature | baseline, 6th months, 12th months, 18th months, 24th months
  Corneal curvature in diopters
non-invasive tear break-up time | 6th months, 12th months, 18th months
  non-invasive tear break-up time in seconds
the lipid layer of the tear film | 6th months, 12th months, 18th months
  the lipid layer of the tear film in nanometers

OTHER OUTCOMES:
ocular surface disease index | baseline, 6th months, 12th months, 18th months, 24th months
  It's a scale for the diagnostic score of dry eye. The total score ranges from 0 to 100, with higher scores indicating more severe symptoms.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Z, Xie R, Luo R, Yao J, Jin L, Zhou Z, Chen K, Zhuo X, Zhu Y, Zhuo Y. Comparisons of Using Cycloplegic Biometry Versus Non-cycloplegic Biometry in the Calculation of the Cycloplegic Refractive Lens Powers. Ophthalmol Ther. 2022 Dec;11(6):2101-2115. doi: 10.1007/s40123-022-00569-w. Epub 2022 Sep 16. PMID 36114405